CLINICAL TRIAL: NCT06305208
Title: A UK Registry for Metabolic and Bariatric Endoscopic Interventions
Acronym: UK-ENDOMAB
Status: Recruiting | Type: Observational
Sponsor: Cleveland Clinic London (Other)
Responsible Party: Sponsor
Other Study IDs: CCLR-23-018
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary bariatric endoscopic procedures
  Interventions: Device: Endoscopic gastric suturing; Device: Endoscopic gastric plication; Device: Intragastric balloon(s)
- Revisional bariatric endoscopic procedures
  Interventions: Device: Revisional gastroplasty; Device: Transoral outlet reduction endoscopy (TORe)
- Primary metabolic endoscopic procedures
  Interventions: Device: Duodenal mucosal resurfacing (DMR)

INTERVENTIONS:
Device: Endoscopic gastric suturing — Endoscopic suturing of the stomach to reduce volume and promote weight loss with either the Apollo Overstitch or Overstitch Sx system.
  Other Names: Endoscopic sleeve gastroplasty (ESG; Apollo Overstitch)
  Groups: Primary bariatric endoscopic procedures
Device: Endoscopic gastric plication — Endoscopic plication of the stomach to reduce volume and promote weight loss with either the POSE or Endomina system.
  Other Names: Primary obesity surgery endoluminal (POSE), Endomina system
  Groups: Primary bariatric endoscopic procedures
Device: Revisional gastroplasty — Endoscopic suturing or plication of the stomach among patients who have previously undergone gastroplasty, sleeve gastrectomy, or Roux-en-Y gastric bypass to restrict the stomach and promote weight loss
  Groups: Revisional bariatric endoscopic procedures
Device: Transoral outlet reduction endoscopy (TORe) — Reduction of the size of the gastro-jejunal anastomosis among patients who have previously undergone Roux-en-Y gastric bypass to promote weight loss. A variety of techniques may be used alone or in isolation including suturing (Apollo Overstitch), plication (POSE), argon photocoagulation, and endoscopic submucosal resection/dissection.
  Groups: Revisional bariatric endoscopic procedures
Device: Duodenal mucosal resurfacing (DMR) — Endoscopic ablation of the post-ampullary duodenal mucosal to enhance improvement in glycaemic control among patients with type 2 diabetes.
  Groups: Primary metabolic endoscopic procedures
Device: Intragastric balloon(s) — The insertion of an intragastric implant into the stomach, which is subsequently filled with air or water to promote weight loss. Several intragastric balloons are available including Allurion, Heliosphere, Obalon, Orbera, and Spatz.
  Groups: Primary bariatric endoscopic procedures

SUMMARY:
In the UK alone, obesity is a major health problem with more than one quarter of adults estimated to be obese. Obesity promotes the development of many serious diseases including diabetes, heart disease, kidney disease, and increased risk of some cancers. Patients living with obesity also suffer from significant symptoms that impact their life including shortness of breath, back pain, poor mobility, and poor mental health. Traditional methods to help lose weight include low calorie diets and increased exercise. These may be effective in the short-term, but due to powerful biological mechanisms they are hard to maintain over the long-term and most individuals are unable to achieve normal weight. This means many people may need bariatric surgery that is highly effective at lowering body weight, but it is associated with complications and not all patients will want or be able to undergo surgery. This has led to the development of many new obesity treatments that are completed with an endoscope. An endoscope is a thin flexible tube that has a camera at the end. It is inserted through the mouth and into the stomach and small bowel. There are various procedures that can be done at the time of endoscopy that have been shown to be effective with a low number of side-effects. These are still relatively new compared to more traditional treatments and only a small number of doctors can perform them within the UK. Due to these limitations, the aim of this registry is to obtain real-world information on the safety and effectiveness of these procedures across the UK. The investigators hope over time this will improve the knowledge of clinicians about treating obesity with endoscopy and support future access and funding to these treatments.

DETAILED DESCRIPTION:
This is a national, multi-centre, prospective, UK registry that aims to determine the safety and efficacy of metabolic and bariatric endoscopic procedures used in the treatment of obesity and related complications. The investigators will do this by determining the effect of primary bariatric procedures (gastroplasty, intragastric balloons (IGB)), revisional bariatric procedures (Transoral outlet reduction endoscopy (TORe), gastroplasty revision), and primary metabolic procedures (Duodenal Mucosal Resurfacing (DMR)), completed by endoscopists within the UK.

The objective of this registry is to collect demographic, procedural and follow-up outcome data on the use of metabolic and bariatric endoscopic procedures in patients with obesity and/or obesity-related complications. This registry will provide real-life outcomes on the use of these novel endoscopic devices from multiple centres participating across the UK to provide longer-term safety and efficacy data. In addition, the registry will enable development of a UK-wide research network to support further research, innovation, and training into metabolic and bariatric endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a primary or revisional bariatric or metabolic endoscopic procedure.
* Age ≥ 18 years old
* Able to give written informed consent.

Exclusion Criteria:

* Any bariatric or metabolic endoscopic procedure performed outside the UK.
* Any bariatric or metabolic endoscopic procedure not currently listed within the registry protocol or agreed by the steering committee.
* Unable to provide written informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients within the United Kingdom (UK) who have, or plan to, undergo a primary or revisional bariatric or metabolic endoscopic procedure for the treatment of obesity or metabolic disease in the UK
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2034-02-01 (Estimated); Study Completion 2039-02-01 (Estimated)

PRIMARY OUTCOMES:
Total body weight loss percentage (TBWL%) | 6-months, 1-, 2-, 3-, 5-years
  For primary or revisional bariatric procedures: Percentage weight loss will be calculated using the following formula: TBWL% = [(weight at the baseline-weight at the end of time period)/weight at baseline] x 100
Change in glycated haemoglobin (HbA1c; mmol/mol) | 6-months, 1-, 2-, 3-, 5-years
  For primary metabolic procedures
Change in the number and dose of anti-diabetic medications | 6-months, 1-, 2-, 3-, 5-years
  For primary metabolic procedures

SECONDARY OUTCOMES:
Procedure time (mins) | Baseline
Inpatient stay (days) | 6-months, 1-, 2-, 3-, 5-years
Adverse events | 30-day, 6-months, 1-, 2-, 3-, 5-years
Change in systolic blood pressure measurements (mmHg) | 6-months, 1-, 2-, 3-, 5-years
Change in diastolic blood pressure measurements (mmHg) | 6-months, 1-, 2-, 3-, 5-years
Changes in number and dose of anti-hypertensive medications (n) | 6-months, 1-, 2-, 3-, 5-years
Changes in low-density lipoprotein cholesterol (mmol/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in triglycerides (mmol/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in high-density lipoprotein cholesterol (mmol/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in total cholesterol (mmol/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in alanine transaminase (IU/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in aspartate aminotransferase (IU/L) | 6-months, 1-, 2-, 3-, 5-years
Changes in Fibrosis-4 Index for Liver Fibrosis | 6-months, 1-, 2-, 3-, 5-years
  The Fibrosis-4 Index for Liver Fibrosis provides a probability score for the presence of hepatic fibrosis. It is based on age, ALT, AST, and platelet count. The range of the score is wide but there are two main cut-offs point for prediction of advanced fibrosis (<1.3 and >2.67). Higher scores indicate a higher likelihood of advanced fibrosis.
Changes in non-alcoholic fatty liver disease fibrosis score | 6-months, 1-, 2-, 3-, 5-years
  The non-alcoholic fatty liver disease fibrosis score provides a probability score for the presence of hepatic fibrosis. It is based on age, body mass index, impaired fasting glucose, ALT, AST, albumin and platelet count. The range of the score is wide but there are two main cut-offs for prediction of advanced fibrosis (<-1.455 and >0.676). Higher scores indicate a higher likelihood of advanced fibrosis.
Changes in weight (kg) | 6-months, 1-, 2-, 3-, 5-years
Changes in body mass index (kg/m2) | 6-months, 1-, 2-, 3-, 5-years
Changes in glycated haemoglobin (HbA1c; mmol/mol) | 6-months, 1-, 2-, 3-, 5-years
Changes in number and dose of anti-diabetic medications (n) | 6-months, 1-, 2-, 3-, 5-years
Changes in number and dose of anti-obesity medications (n) | 6-months, 1-, 2-, 3-, 5-years
Changes in health-related quality of life scores (EuroQol-5D-5L) | 6-months, 1-, 2-, 3-, 5-years
  The EuroQol-5D-5L is a quality of life questionnaire that is composed of five questions scored 1-5 that do not have an arithmetic value and a visual analogue scale between 0-100. Participants are simply given a five digit code (e.g. 13455) and a visual analogue score (e.g. 78), which can then be interpreted through reference value sets in the corresponding country.

CONTACTS AND LOCATIONS:
Overall Officials: Rehan Haidry, MD, Principal Investigator — Cleveland Clinic London
Locations (1):
- Cleveland Clinic London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No